CLINICAL TRIAL: NCT05732675
Title: Building Resilience to Minority Stress and HIV-related Stigma for Promoting Positive Sexual Health Among Vietnamese High-risk Men
Brief Title: Stress and HIV-related Stigma Among Men in Viet Nam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: The Center for Applied Research for Men and Community Health (Unknown)
Responsible Party: Principal Investigator, Frankie Wong, McKenzie Endowed Professor of Health Equity Research, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REL00000085
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2023-03

CONDITIONS: Bisexuality; Homosexuality; HIV Infections
MeSH Terms: conditions — Bisexuality; Homosexuality; HIV Infections

STUDY DESIGN:
Intervention Model Description: This study follows a parallel design, where participants are randomized into two arms-immediate intervention and waitlist control. The study aims to test the feasibility and efficacy of the ESTEEM intervention in small groups, with ongoing assessment over a 6-month period.
Masking Description: This study does not involve masking of participants, care providers, or investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention (Other): Participants immediately enter the intervention upon enrollment
  Interventions: Behavioral: "Vina-STEAM" (Skills to Empower Affirmative Men)
- Waitlist (Other): Participants enter a waitlist for 4-weeks prior to participating in the intervention
  Interventions: Behavioral: "Vina-STEAM" (Skills to Empower Affirmative Men)

INTERVENTIONS:
Behavioral: "Vina-STEAM" (Skills to Empower Affirmative Men) — The investigators propose and pilot test a community-based, peer-driven minority stress as well as HIV-stigma reduction program in small group of GBM in Ho Chi Minh City, Viet Nam.

SUMMARY:
Participants are Vietnamese national. Over the course of the study activities, approximately 184 self-identified Vietnamese national gay and bisexual men ages 18 and above living in HCMC, Viet Nam, as well as 10 key informants (about 5 females) ages 18 and above will participate in the study.

DETAILED DESCRIPTION:
The mixed-method study will involve: (1) preparation stage; (2) formative stage, where qualitative data from Vietnamese GBM and key informants will inform the adaptation of the ESTEEM package; (3) feasibility test, where the adapted intervention will be piloted-test in a small sample (4 small group, N = 24) of GBM and further adjusted on the pilot-test results; and (4) small-scale efficacy test of the adjusted intervention using a randomized waitlist controlled design in a cohort of 120 GBM, where they will be randomly assigned to either the immediate intervention (6 groups) or a waitlist arm (6 groups) with 10 men per groups. During the preparation stage, the investigators will obtain ethical approval from the Florida State University's Institutional Review Board. The investigators will identify and hire staff knowledgeable about the local socio-cultural context pertaining to GBM, fluent in Vietnamese, and familiar with research-oriented studies. All personnel and individual contacting with the study on human participants will be trained on human subject protection. During the qualitative formative stage, the investigators will conduct individual interviews (N = 15) of GBM community representatives, focus group (4 group, N = 25) with GBN community representative and individual interviews (N = 10) of key informants. Key informants (e.g., outreach workers, counselors, consultant, psychologists, program managers) will consist of adults with experience working with GBM in the areas of mental or sexual health, stigma, and/or legal protection. Interviews and focus groups will be audio-recorded. The investigators will intersperse key informant interviews, individual interviews, and focus groups with GBM and the process of ESTEEM adaptation in an iterative manner. For the feasibility test stage, the investigators will recruit 24 GBM to pilot test the adapted intervention in small groups (N = 6 per group) setting to meet once weekly for a period of 8 week. During the intervention, qualitative data will be collected via baseline and endline surveys. Qualitative data will be collected from individual interviews after each individual session in addition to ta final individual and 4 focus groups after completion of all sessions in the intervention. These data will be used to revise the intervention as needed for the small-scale efficacy stage. Audio-recordings of interviews and focus groups from the formative and feasibility test stages will be transcribed verbatim and analyzed in MaxQDA software using thematic analysis. Data from interviews and focus groups will be complemented by information from peer facilitators' oral feedback and participants' open-ended questionnaires.

Qualitative data analysis will be guided by the intervention feasibility domains --acceptability, demand, implementation, practicality, adaptation, integration, and expansion. Due to the small sample size (N = 24) in the feasibility test no inferential statistical analysis of quantitative data will be performed. The investigators will only determine the direction of changes in the primary outcomes and assess effect sizes. For the small-scale efficacy stage, the investigators will enroll and assign 120 consented participants to 12 small groups and with 10 individuals in each group. Then the investigators will randomize the small groups into the immediate intervention and waitlist arms (6 groups in each arm). All participants will complete 3 waves of data collection: baseline, 3-month follow-up, and 6-month follow-up. Power calculations (using PROC POWRR in SAS 9.4 and assuming an intra-cluster correlation of 10%) demonstrates that a sample size of 120 is sufficiently large to detect medium effect size of d = 0.477 via a one-sided independent t-test. The investigators will include all randomized participants into the analysis using an intent-to-treat approach. The investigators will use mixed models with appropriate distribution and link functions based on endpoint variable properties along with repeated measures approach to account for within individual and group correction.

ELIGIBILITY:
Inclusion Criteria:

* born as a biological male and self-identifying as a man
* ages 18 and above,
* self-reported as gay or bisexual
* a verifiable HIV-negative status
* reporting at least one episode of unprotected anal sex with a casual male partner or male partner with positive or unknown HIV-status in the past 30 days
* able and willing to provide verbal and written informed consent in Vietnamese
* intending to Stay in Ho Chi Minh City, Viet Nam, not to leave the city for more than one week in the next two months.

Exclusion Criteria:

* Has a known psychiatric disorder
* is under influence of alcohol and/or drugs
* ages 17 and below.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Increase in HIV testing. | 24 months
  Increase in HIV testing

CONTACTS AND LOCATIONS:
Overall Officials: Frankie Wong, Principal Investigator — Florida State University
Locations (1):
- Center for Research for Men and Gender Health, Ho Chi Minh City, Vietnam